CLINICAL TRIAL: NCT00631566
Title: Prospective Study on the Incidence, Predictors, and Characteristics of Methicillin-Resistant Staphylococcus Aureus Infections and a Randomized, Double-Blind Study on Decolonization Procedures for Prevention of MRSA Infections Among HIV-Infected Persons
Brief Title: Prospective Study of Methicillin-Resistant Staphylococcus Aureus (MRSA) Among HIV-Infected Persons
Acronym: MRSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); US Military HIV Research Program (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCRP-003-RV210
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; Staphylococcal Infections
Keywords: HIV; Methicillin-resistant Staphylococcus aureus (MRSA); HIV and Staphylococcus aureus infection
MeSH Terms: conditions — HIV Infections; Staphylococcal Infections | interventions — Mupirocin; Hexachlorophene; Triclosan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Mupirocin (Bactroban) 2%; hexachlorophene (pHisoHex) 3%
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- No MRSA colonization (No Intervention)

INTERVENTIONS:
Drug: Mupirocin (Bactroban) 2%; hexachlorophene (pHisoHex) 3% — BACTROBAN NASAL is a white to off-white ointment that contains 2.15% w/w mupirocin calcium (equivalent to 2.0% pure mupirocin free acid) in a soft white ointment base. The inactive ingredients are paraffin and a mixture of glycerin esters (SOFTISAN 649).
  pHisoHex, brand of hexachlorophene detergent cleanser, is an antibacterial sudsing emulsion for topical administration.
  Some randomized patients will receive mupirocin (Bactroban) nasal ointment plus hexachlorophene (pHisoHex) body washes for seven days.
  Arms: 1
Drug: Placebo — Some randomized patients will receive a placebo nasal ointment (white petroleum) and a placebo body soap with no antimicrobial activity for seven days.
  Arms: 2

SUMMARY:
This study will prospectively evaluate the prevalence and incidence (over a two year period) of MRSA colonization and infection among HIV-infected military beneficiaries to determine predictors for the development of MRSA colonization and infection. This study will also investigate the utility of decolonization procedures for clearance of MRSA carriage and prevention of MRSA infections. Finally, the molecular characteristics and the antimicrobial sensitivities of isolates in this population will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years of age) who are HIV positive by a reactive screening (ELISA, EIA) and a confirmatory test (Western blot) and who are able to attend the study visits which are every 6 months (+/- 2 months), at the minimum

Exclusion Criteria:

* Known allergy to mupirocin (Bactroban®) nasal ointment or hexachlorophene (pHisoHex®) soaps or constituents of these products.
* Age less than 18 years.
* Inability to remain in the study for the two year duration.
* Pregnant or breastfeeding females.
* Females who intend to become pregnant during the two year study time period.
* Persons who are healthcare providers with direct patient contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2007-05; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Naval Medical Center San Diego/Infectious Disease Division, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - San Antonio Military Medical Center (BAMC/WHMC), San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

REFERENCES:
- [Background] Vyas KJ, Shadyab AH, Lin CD, Crum-Cianflone NF. Trends and factors associated with initial and recurrent methicillin-resistant Staphylococcus aureus (MRSA) skin and soft-tissue infections among HIV-infected persons: an 18-year study. J Int Assoc Provid AIDS Care. 2014 May-Jun;13(3):206-13. doi: 10.1177/2325957412473780. Epub 2013 Apr 19. PMID 23603632
- [Result] Crum-Cianflone NF, Shadyab AH, Weintrob A, Hospenthal DR, Lalani T, Collins G, Mask A, Mende K, Brodine SK, Agan BK; Infectious Disease Clinical Research Program HIV Working Group. Association of methicillin-resistant Staphylococcus aureus (MRSA) colonization with high-risk sexual behaviors in persons infected with human immunodeficiency virus (HIV). Medicine (Baltimore). 2011 Nov;90(6):379-389. doi: 10.1097/MD.0b013e318238dc2c. PMID 22033452
- [Result] Weintrob A, Bebu I, Agan B, Diem A, Johnson E, Lalani T, Wang X, Bavaro M, Ellis M, Mende K, Crum-Cianflone N. Randomized, Double-Blind, Placebo-Controlled Study on Decolonization Procedures for Methicillin-Resistant Staphylococcus aureus (MRSA) among HIV-Infected Adults. PLoS One. 2015 May 27;10(5):e0128071. doi: 10.1371/journal.pone.0128071. eCollection 2015. PMID 26018036
- [Result] Crum-Cianflone NF, Wang X, Weintrob A, Lalani T, Bavaro M, Okulicz JF, Mende K, Ellis M, Agan BK. Specific Behaviors Predict Staphylococcus aureus Colonization and Skin and Soft Tissue Infections Among Human Immunodeficiency Virus-Infected Persons. Open Forum Infect Dis. 2015 Mar 6;2(2):ofv034. doi: 10.1093/ofid/ofv034. eCollection 2015 Apr. PMID 26380335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected adults from four US Military HIV clinics were prospectively enrolled during routine visits. Enrollment occurred between May 2007 and May 2010 and follow-up visits were conducted until August 2012.
Groups:
- Mupirocin/Hexachlorophene Group: Participants with MRSA colonization who were randomized to receive:
  Mupirocin (Bactroban) 2%; hexachlorophene (pHisoHex) 3%: BACTROBAN NASAL is a white to off-white ointment that contains 2.15% w/w mupirocin calcium (equivalent to 2.0% pure mupirocin free acid) in a soft white ointment base. The inactive ingredients are paraffin and a mixture of glycerin esters (SOFTISAN 649).
  pHisoHex, brand of hexachlorophene detergent cleanser, is an antibacterial sudsing emulsion for topical administration.
  Some randomized patients will receive mupirocin (Bactroban) nasal ointment plus hexachlorophene (pHisoHex) body washes for seven days.
- Placebo Group: Participants with MRSA colonization who were randomized to receive:
  Placebo: Some randomized patients will receive a placebo nasal ointment (white petroleum) and a placebo body soap with no antimicrobial activity for seven days.
- No MRSA Colonization: Patients who did not have any MRSA colonization.
Period: Overall Study
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization
Started | 21 | 28 | 501
Completed | 19 | 24 | 501
Not Completed | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization | Total
Number analyzed (Participants) | 21 | 28 | 501 | 550
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [34 to 47] | 46 [38 to 52] | 42 [32 to 49] | 42 [33 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 36 | 37
  Male | 20 | 28 | 465 | 513
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9 | 15 | 287 | 311
  African-American | 10 | 12 | 174 | 196
  Other | 2 | 1 | 40 | 43
Region of Enrollment [Number; unit: participants]
  United States | 21 | 28 | 501 | 550
Current CD4 count [Median (Inter-Quartile Range); unit: cells/mm3] | 494 [312 to 695] | 500 [424 to 618] | 534 [404 to 706] | 529 [402 to 704]
CD4 by category [Count of Participants; unit: Participants]
  <350 cells/mm3 | 7 | 2 | 93 | 102
  350-499 cells/mm3 | 4 | 12 | 117 | 133
  >/= 500 cells/mm3 | 10 | 14 | 290 | 314

OUTCOME MEASURES:

1. Primary Outcome: The Presence of MRSA on Repeated Swabs to Assess the Efficacy of These Medications on Clearing MRSA Colonization
Description: MRSA colonization at 6-months post-randomization
Time Frame: 6 months
Population: Only 80% of the 49 initial randomizations had 6-month colonization data and were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization
Number analyzed (Participants) | 18 | 21 | 501
Participants | 12 | 14 | 0

2. Secondary Outcome: To Determine the Prevalence and Incidence of MRSA Colonization of the Nares, Throat, Perirectal, Axilla, and Groin Areas Among HIV Infected Patients and to Study Changes in the Colonization Rates Over Time.
Time Frame: Every 6 months
Population: Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization
Number analyzed (Participants) | 21 | 28 | 501
Participants
  Nares | 17 | 18 | 0
  Throat | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | 0
  Perirectal | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | 0
  Groin | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | 0
  Axilla | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | NA — Due to small numbers, the colonization in the sites other than nares, the counts were not further identified between the treatment group and the placebo group. | 0

3. Secondary Outcome: To Evaluate the Change in CD4 Counts and HIV Viral Loads During the Time of a MRSA or Soft Tissue Infection.
Description: This outcome measure was not analyzed/reported due to resource limitations.
Time Frame: At time of infection
Population: As requested, the number of participants was set to zero since this analysis was not conducted.
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: To Characterize the Molecular Characteristics and the Antimicrobial Sensitivities of MRSA Isolates in This Population.
Description: This outcome measure was not analyzed/reported due to resource limitation.
Time Frame: at time of positive MRSA results
Population: As requested, the number of participants was set to zero since this analysis was not conducted.
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years following enrollment into the study
Arm/Group | Mupirocin/Hexachlorophene Group | Placebo Group | No MRSA Colonization
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/28 | 0/501
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/28 | 0/501
Other Adverse Events (participants affected / at risk) | 0/21 | 0/28 | 0/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mupirocin/Hexachlorophene Group (N=21) | Placebo Group (N=28) | No MRSA Colonization (N=501)
Hospitalization for gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Low rates of MRSA infections and SSTI during follow-up. Mostly males. Data for counts by arm other than nares for Outcome #2 are estimates from proportions and overall sample as these data were not available when record completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT00631566/Prot_SAP_000.pdf